CLINICAL TRIAL: NCT01744301
Title: A Cohort Study With a Nested Case Control Analysis on the Association Between Acid-suppressing Drugs and Seizures Using THIN Database in the UK
Brief Title: Acid Suppressing Drug Seizure Epidemiology Study
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9612N00017
Record Dates: First submitted 2012-12-05; First posted 2012-12-06 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2015-12

CONDITIONS: Seizure
Keywords: Seizure; Acid-suppressing drugs; Epidemiology
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- All patients newly prescribed PPI: All patients newly prescribed PPI
  Interventions: Drug: Risk of seizure
- All patients newly prescribed H2RA: All patients newly prescribed H2RA
  Interventions: Drug: Risk of seizure

INTERVENTIONS:
Drug: Risk of seizure — Patients newly prescribed PPI and H2RA, respectively

SUMMARY:
The purpose of this study is

1. to estimate the incidence of seizure in the general population and stratified by epilepsy status
2. To estimate the relative risk of seizure associated with use of proton pump inhibitors and histamine 2 receptor antagonist and stratified by epilepsy status

DETAILED DESCRIPTION:
A cohort study with a nested case control analysis on the association between acid-suppressing drugs and seizures using THIN database in the UK

ELIGIBILITY:
Inclusion Criteria:

* Primary care physician for at least 2 years.
* Computerized prescription history of at least 1 year.
* Patients will have to be free of acid-suppressing drugs (PPI or H2RA) for at least one year.
* No diagnosis of cancer.
* No alcohol abuse or alcohol-related disease- No drug abuse.

Exclusion Criteria:

* Patients with at least 1 prescription of PPI or H2RA in the year prior to start date.
* Cancer before start date.
* Alcohol abuse or alcohol-related disease before start date.
* Drug abuse before start date.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals aged 20-84 years from 1 January 2005 to 31 December 2011, who have been enrolled with their primary care physician for at least 2 years and have a computerized prescription history of at least 1 year. Patients will have to be free of acid-suppressing drugs (PPI or H2RA) for at least one year, and never have a diagnosis of cancer, alcohol abuse or alcohol-related disease, or drug abuse.
Sampling Method: Non-Probability Sample
Enrollment: 8605 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence of seizure in the general population and stratified by epilepsy status. | Participants will be followed for the duration of the study period 1 January 2005-31 December 2011, an expected average of 3 years.
Follow-up of safety outcomes: First recorded entry of seizure. | Participants will be followed for the duration of the study period 1 January 2005-31 December 2011, an expected average of 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Luis a Garcia Rodriguez, MD, Principal Investigator — CEIFE (Centro Espanol de Investigacion Farmacoepidemiologica - Spanish Centre for Pharmacoepidemiologic Research )
Locations (1):
- Research Site, Madrid, Spain

REFERENCES:
- [Background] Saez ME, Gonzalez-Perez A, Gaist D, Johansson S, Nagy P, Garcia Rodriguez LA. Risk of seizure associated with use of acid-suppressive drugs: An observational cohort study. Epilepsy Behav. 2016 Sep;62:72-80. doi: 10.1016/j.yebeh.2016.06.039. Epub 2016 Jul 21. PMID 27450309
- Available data/document: Study Protocol: CSR Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7112&studyid=674&filename=D9612N00017_Seizure_Study_report_synopsis_FINAL_redacted.pdf — D9612N00017_Seizure_Study_report_synopsis_FINAL_redacted